CLINICAL TRIAL: NCT04728126
Title: Menopausal Symptoms and Burnout: Comparison of Occupational Health Issue Among Health Professionals in University Hospitals of UMC in Nur-Sultan
Brief Title: Menopausal Symptoms and Burnout: Comparison of Occupational Health Issue Among Health Professionals in UMC Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nazarbayev University Medical Center (Other)
Collaborators: University of South Florida (Other); Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Sanja Terzic, Principal Investigator, Nazarbayev University Medical Center
Organization: Nazarbayev University (Other)
Other Study IDs: 023-2020
Record Dates: First submitted 2021-01-22; First posted 2021-01-28 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Menopause; Burnout Syndrome
Keywords: Menopause; Quality of life; Quality of work life; Burnout; Emotional exhaustion
MeSH Terms: conditions — Burnout, Psychological; Emotional Exhaustion | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Female health-care givers aged 45 to 64 years. The study participants will be recruited from UMC (Clinical Academic Department (CAD) of Women's Health, Pediatric Clinical Academic Department, Republic Diagnostic Center (RDC) and National Center for Children's Rehabilitation (NCCR)), Nur-Sultan, Kazakhstan.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The questionnaire will include socio-demographic information (i.e., gender, age, job seniority) and sub-scales for measuring study variables (i.e., menopausal symptoms, social and personal resources, burnout, and work ability).
  Menopausal symptoms will be assessed using the Menopause-Specific Quality of Life questionnaire.
  Job burnout will be measured through OBI inventory, which consists of 16 items describing the states of emotional exhaustion and detachment - two core dimension of burnout, and were developed to meet different occupational groups.
  The menopause and the quality of working environment will be assessed using the Questionnaire developed by National Health Service in England and Wales.

SUMMARY:
This study aims at evaluating the burnout in women healthcare providers (physicians and nurses) Kazakhstan settings, and to investigate the potential parameters that play a role in increasing the risk of burnout. This study would apply the Oldenburg Burnout Inventory (OBI) in a sample of menopausal healthcare providers belonging to the University Medical Center (UMC) - quaternary healthcare institution in Nur-Sultan, Kazakhstan.

DETAILED DESCRIPTION:
Menopause is a complex physiological process that marks the end of the reproductive phase of a woman's life, and some women in that population refer to various symptoms like hot flashes, sleep disturbances, decreased physical strength, mood changes, and bladder irritability. The increasing presence of women in the workplace and the aging of the women's workforce have elicited growing interest in the link between menopause and work. Studies in the occupational-medicine field provide evidence of how certain aspects of the physical work environment exacerbate menopausal symptoms. Furthermore, there are direct and indirect costs from a lack of organizational support for menopausal women in terms of increased absenteeism, presenteeism, and medical checkups.

Occupational Burnout (OB) is a syndrome of physical and psychological exhaustion of health care professionals. It has three dimensions relating to emotional exhaustion, depersonalization and lack of personal achievements. Extant studies in the occupational health psychology (OHP) field have highlighted many factors in the health-care providers work environment that might increase the risk of developing burnout. It has been well-established that among human-service professionals, the most important burnout risk is represented by the emotionally demanding relationships between caregivers and recipients.

Excessive workload and loss of control in one's profession are cited as the top reasons for burnout among physicians. Likewise, among surgeons, a primary contributing factor for burnout is long working hours, with only a third of surgeons feeling their work schedule had left enough time for personal or family life. Work family conflicts are also more common if surgeons are married to another physician or surgeon. Clearly these reasons imply that a primary root of the problem lies with organizations and care delivery systems rather than the individuals. Furthermore, workplace politics can be associated with a higher risk of burnout, depression and coronary artery disease. Adequate staffing, good leadership and support were found to reduce the risk of burnout, highlighting the importance of fair hospital management, policy and practice. Nevertheless, causes of burnout are not always organizational in nature; a proportion are due to the mishandling of stress related to the profession or at work. This is especially evident among vulnerable physicians with traits including idealism, perfectionism and a great sense of responsibility. Early career physicians (i.e. ≤ 5 years in practice) who have these personality traits are at a greater risk, particularly during the first few years immediately after completion of their fellowship. An early presence in academic and private settings and being involved in interventional procedures can be stressful to an early career physician. In addition, certain patient factors may also contribute to burnout; these include unrealistic expectations, declining patient health and aggression from patients. Prolonged patient contact and development of family-like relationships may also result in emotional detachment and burnout.

In summary, contributing factors leading to burnout are poor working conditions with long work shifts, stressful on-call duties, lack of appreciation, and poor social interactions. Burnout can lead to adverse consequences, such as depression, substance use, and suicidal ideation. This can result in poor patient care, increasing total length of stay, re-admissions, and major medical errors. Due to increased scrutiny of patient and healthcare costs, along with increased lawsuits as a result of major medical errors, it is crucial for both the hospital management and healthcare providers to recognize and address burnout. Comprehensive professional training such as Cognitive behavioral therapy (CBT), stress-reducing activities such as mindfulness and group activities, and strict implementation of work-hour limitations are a few methods that may help to manage burnout and increase productivity in hospitals.This study aims at evaluating the burnout in women healthcare providers (physicians and nurses) Kazakhstan settings, and to investigate the potential parameters that play a role in increasing the risk of burnout. This study would apply the OBI in a sample of menopausal healthcare providers belonging to the UMC - quaternary healthcare institution in Nur-Sultan, Kazakhstan.

ELIGIBILITY:
Inclusion Criteria:

* menopause

Exclusion Criteria:

* severe chronic diseases, including psychological/psychiatric comorbidities and use of specific drugs for them

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Since this study is aimed to investigate and determine the quality of life in menopausal women, the participants are menopausal women aged 45 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Menopause Quality of Life Measurement | 36 month
  Participants will be asked to fill a self-administered Menopause-Specific Quality of Life questionnaire, which comprises 29 items.
  This Menopause-Specific Quality of Life contains items that assess 4 main types of menopausal symptoms: vasomotor, psychosocial, physical, sexual. Each item is rated as present or not present; if present, how bothersome the items are on a scale of 0 (not bothersome) to 6 (extremely bothersome).
Job burnout | 36 month
  Job burnout will be measured using Oldenburg Burnout Inventory.
  Oldenburg Burnout Inventory consists of 16 items on the states of emotional exhaustion and detachment, and were developed to meet different occupational groups. The degree of agreement with 16 items of Oldenburg Burnout Inventory uses scale from 1 to 4, where 1- strongly agree and 4 - strongly disagree.
The menopause and quality of working environment | 36 month
  The menopause and quality of working environment will be assessed using a questionnaire developed by National Health Service in England and Wales.
  This questionnaire will enable information about the menopause experience, how menopause affects the workplace and vice versa. Moreover, it will provide information about the performance management during menopause and enable foundations about the eventual need for possible ways of raising awareness at work.

CONTACTS AND LOCATIONS:
Overall Officials: Milan Terzic, Study Director — Nazarbayev University Medical Center; Gauri Bapayeva, Study Director — Nazarbayev University Medical Center